CLINICAL TRIAL: NCT06757517
Title: Effects of Intranasal Oxytocin in the Treatment of Benzodiazepine Withdrawal: A Pilot Randomized Parallell Group Placebo-Controlled Trial
Brief Title: Effects of Intranasal Oxytocin in the Treatment of Benzodiazepine Withdrawal: A Pilot RCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Lade Behandlingssenter, Blå Kors (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 32672
Record Dates: First submitted 2024-10-17; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Benzodiazepine Dependence
Keywords: intranasal oxytocin; oxytocin; benzodiazepines; benzodiazepine dependence; benzodiazepine withdrawal
MeSH Terms: interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants in the placebo arm will receive a saline solution. Saline is an inert substance, meaning it has no therapeutic effect, making it an ideal placebo. The saline solution will be administered in the same manner as the experimental treatment. The treatment is administered intranasally. The treatment is blinded. Neither the participants nor the researchers know who is receiving the placebo and who is receiving the active treatment. Participants in the placebo arm will be monitored the same as those in the treatment arm. Participants will be fully informed about the possibility of receiving a placebo and will provide informed consent. The same outcome measures will be used for both the placebo and treatment arms.
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)
- Oxytocin (Experimental): Participants in this arm will receive intranasal oxytocin. The dosage and administration schedule will be consistent with the study protocol. Participants will receive 48 international units (IU) of oxytocin. The oxytocin will be administered intranasally using a nasal spray. Participants will insert the nasal spray container approximately 1 cm into each nostril and spray. They will wait 15 seconds before repeating administration until they have received a total of 4 puffs (2 in each nostril) per session thrice daily.
  Interventions: Drug: Oxytocin nasal spray

INTERVENTIONS:
Drug: Oxytocin nasal spray — Syntocinon contains synthetic oxytocinfor intranasal use, 6.7 microg (4 IU) per dose. We are planning to use 4 insufflations (16 IU) three times daily (i.e. a total daily dose of 48 IU).
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Saline (NaCl 0,9 %) (placebo) — Saline intranasal placebo comparator
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if oxytocin administered as a nasal spray will reduce withdrawal symptoms in adults during benzodiazepine tapering for 21 days. It will also learn about the safety of oxytocin. The main question it aims to answer are:

Does oxytocin reduce benzodiazepine withdrawal symptoms and make it easier to succeed tapering? Does oxytocin help reduce sleep difficulties and anxiety or restlessness during benzodiazepine tapering? Does oxytocin help reduce benzodiazepine craving?

We will compare oxytocin nasal spray to a placebo nasal spray containing regular saline to see if oxytocin works accordingly.

Participants will:

Take oxytocin or a placebo nasalspray, thrice daily for 21 days during inpatient benzodiazepine tapering.

Fill out an online questionnaire every day and keep a record of their symptoms.

DETAILED DESCRIPTION:
Background Benzodiazepine withdrawal can be challenging, often accompanied by severe anxiety, insomnia, and other withdrawal symptoms. Recent studies suggest that intranasal oxytocin (OT) may have anxiolytic properties and could potentially ease withdrawal symptoms. This pilot study aims to evaluate the efficacy and safety of intranasal OT in the treatment of benzodiazepine withdrawal.

Objectives The primary objective is to evaluate if intranasal OT can reduce withdrawal symptoms in patients during benzodiazepine tapering. Secondary objectives include evaluating the safety and tolerability of intranasal OT and its impact on anxiety levels and sleep quality.

Methods

* Design: This is a randomized, parallel-group, placebo-controlled trial.
* Participants: 60 adults (aged 18-65) who are undergoing benzodiazepine tapering.
* Intervention: Participants will be randomly assigned to receive either intranasal OT (24 IU) or a placebo, administered twice daily for four weeks.
* Assessments: Withdrawal symptoms will be measured using the Clinical Institute Withdrawal Assessment for Benzodiazepines (CIWA-B) scale. Anxiety levels will be assessed using the Hamilton Anxiety Rating Scale (HAM-A), and sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI) and actigraphy recordings.

Procedure

1. Screening: Eligible participants will undergo a screening process, including medical history, physical examination, and baseline assessments.
2. Randomization: Participants will be randomly assigned to the OT or placebo group.
3. Treatment Phase: Participants will self-administer the nasal spray thrice daily for three weeks. Participants will fill out daily questionnaires to monitor symptoms and side effects. Weekly urine- and blood samples will be collected.
4. Post-Treatment Follow-Up: Participants will be assessed at the end of the treatment period and again four and twelve weeks post-treatment to evaluate the persistence of effects.

Expected Outcomes It is hypothesized that participants receiving intranasal OT will experience a significant reduction in withdrawal symptoms compared to the placebo group. Improvements in anxiety levels and sleep quality are also anticipated.

Significance This study could provide preliminary evidence for the use of intranasal OT as a supportive treatment for benzodiazepine withdrawal, potentially improving patient outcomes and comfort during the tapering process.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 65 years, taking benzodiazepines at a daily dose of 20-80 mg diazepam-equivalent, and requiring inpatient benzodiazepine withdrawal. Included patients must consent to participate in the study.

Exclusion Criteria:

* Female patients will be excluded if they are pregnant or are planning to become so, or if they are breast-feeding. Individuals incapable of completing questionnaires or giving informed consent will be excluded. Patients with concurrent acute medical or psychiatric illness requiring acute care hospitalization, misuse or dependency of alcohol or pregabalin/gabapentin will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Benzodiazepine withdrawal symptoms | 21 days
  Benzodiazepine withdrawal symptoms severity is measured with CIWA-B score, a 20-item scale where each item can be assigned a score from 0 to 4, i.e. the total score can range from 0 and 80 points. CIWA-B score will be measured daily from baseline (i.e. the day before the intervention starts) to day 21.

SECONDARY OUTCOMES:
Benzodiazepine craving | 21 days
  To test whether there is a difference between oxytocin and placebo on cravings. Comparing cravings scores measured daily with a 6-item Likert scale where the score can range between 0 to 5 points between the two study groups from baseline to day 21. Specifically, the change in scores from baseline to day 21 will compared between the two groups.
Benzodiazepine anxiety and depression symptoms | 21 days
  To test whether there is a difference between oxytocin and placebo on rebound anxiety and depression symptoms. Comparing Hospital Anxiety and Depression rating scale (HAD) scores measuring psychological distress, anxiety and depression between the two study groups measured weekly from baseline to day 21. Specifically, the change in scores from baseline to day 21 will compared between the two groups.
Benzodiazepine sleep distress | 21 days
  To test whether there is a difference between oxytocin and placebo on sleep. Comparing Insomnia Severity Index (ISI) scores measuring sleep difficulties, and sleep variables assessed by actigraphy and Somnofy, between the two study groups from baseline to day 21 during intervention.
Benzodiazepine tapering "freezes" | 21 days
  To test whether there is a difference between oxytocin and placebo in the number of "freezes" in diazepam tapering. A "freeze" (not reducing the diazepam dose as scheduled during tapering) will be noted for each subject and compared between the two study groups.

OTHER OUTCOMES:
Follow-up: Relapse | 15 weeks
  To test whether there is a difference between oxytocin and placebo in time to first benzodiazepine intake (up to 12 weeks after discharge). Comparing time (number of days) to first self-reported benzodiazepine intake after discharge (week 3) between the two study groups, by registration on the follow-up visits at week 7 and week 15.
Follow-up: Benzodiazepine withdrawal symptoms | 15 weeks
  Difference between oxytocin and placebo group on withdrawal symptoms measured with CIWA-B at week 7 and week 15 after discharge.
Follow-up: Benzodiazepine craving | 15 weeks
  To test whether there is a difference between oxytocin and placebo on cravings. Comparing cravings scores measured at week 7 and week 15 after discharge with a 6-item Likert scale where the score can range between 0 to 5 points between the two study groups from baseline to day 21.
Follow-up: Benzodiazepine anxiety and depression symptoms | 15 weeks
  To test whether there is a difference between oxytocin and placebo on rebound anxiety and depression symptoms at week 7 and week 15 after discharge. Comparing Hospital Anxiety and Depression rating scale (HAD) scores measuring psychological distress, anxiety and depression between the two study groups.
Follow-up: Benzodiazepine sleep distress | 15 weeks
  To test whether there is a difference between oxytocin and placebo on sleep distress at week 7 and week 15 after discharge. Comparing Insomnia Severity Index (ISI) scores measuring sleep difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Tone Aurora Pleym, MD, PhD-candidate, Study Chair — NTNU, Blue Cross, Clinic Lade, St. Olavs hospital
Locations (1):
- Blue Cross, Clinic Lade, Trondheim, Trøndelag, Norway